CLINICAL TRIAL: NCT07171255
Title: Improving Exercise Adherence With App Technology for At-Risk Adults Living in Rural Kansas and Nebraska
Acronym: RemoteEx+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005493
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Middle Age and Older Aged Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RemoteEx+ Program (Experimental)
  Interventions: Behavioral: RemoteEx+ Programming

INTERVENTIONS:
Behavioral: RemoteEx+ Programming — The exercise program will include video instruction for all exercises, motivational cues, and ADRD risk education throughout the 16-week exercise program to encourage exercise adherence. RemoteEx+ is optimized to enhance exercise knowledge surrounding dementia risk factors to facilitate ADRD risk reduction and overall health improvement. The purpose of this study is to investigate the efficacy of RemoteEx+ on health outcomes associated with dementia risk in underactive rural adults.

SUMMARY:
Alzheimer's disease and related dementias are a public health crisis impacting individuals across the world. In the United States, adults living in rural areas face an elevated risk for cognitive impairment mainly due to disparities in care, higher sedentary behavior, and reduced education. This project proposes to assess the impact of a remotely delivered exercise program (i.e., RemoteEx+) through a smartphone application. The app is programmed by our team and provides video demonstrations of exercises, workout regimes, motivational messaging, and weekly ADRD risk reduction education. The project aims to assess with a pre/post design the following aims:

* Aim 1. Assess the RemoteEx+ intervention exercise adherence, efficacy, enjoyment, and quality of life. We hypothesize that rural adults will report high exercise adherence (80% of session adherence), efficacy (>50% on Self Efficacy for Exercise), and enjoyment (>5.0 on Intrinsic Motivation Inventory - Interest / Enjoyment Subscale) and that these variables will be positively correlated with quality of life scores (36-Item Short Form Health Survey [SF-36])
* Aim 2. Determine the impact of a technology-driven exercise program on blood pressure and functional mobility associated with dementia risk. We hypothesize that the exercise program will result in improvements in blood pressure and functional mobility (2-minute step test and 30-second chair rise test) and that participants with high exercise adherence will see the greatest improvements in biomarkers associated with reduced dementia risk.
* Aim 3. Reduce health disparities among rural-dwelling Nebraska and Kansas residents. We hypothesize that RemoteEx+ will reduce barriers to exercise (Barriers to Being Active Quiz and improve knowledge surrounding dementia and modifiable risk factors (Dementia Knowledge Assessment Tool - Version 2 [DKAT2]) that will result in fewer lifestyle-related health disparities for the communities involved in this study.

The results from this project will inform whether RemoteEx+ has an impact on the stated outcomes above for adults living in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years
* Characterized as underactive by the Telephone Assessment of Physical Activity (TAPA)50
* Self-reported proficiency in English
* Own a smartphone and willing to download an application
* Primary care provider clearance to participate for those who do not pass the PAR-Q+51
* Live in a rural area (Rural-Urban Commuting Area [RUCA] Codes) 52

Exclusion Criteria:

* Contraindications to high-intensity exercise
* Cognitive impairment (<19 on the Telephone Montreal Cognitive Assessment [MoCA])
* Neurodegenerative or acute neurological diagnoses (e.g., Parkinson's disease, stroke, traumatic brain injury)
* Orthopedic surgery or injuries in the last 6 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Baseline and Week 16

SECONDARY OUTCOMES:
Cardiovascular Endurance | Baseline and Week 16
  2-Minute Step Test
Lower Extremity Strength | Baseline and Week 16
  30-second chair rise test
Exercise Adherence | Baseline and Week 16
  % of sessions completed over the 16-week program
Exercise Efficacy | Baseline and Week 16
  Self Efficacy for Exercise (SEE) Scale (points)
Quality of Life Improvement | Baseline and Week 16
  36-Item Short Form Health Survey
Barriers to Being Active | Baseline and Week 16
  Barriers to Being Active Quiz
Knowledge of dementia | Baseline and Week 16
  Dementia Knowledge Assessment Tool

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emporia State University, Emporia, Kansas
  - Creighton University, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided